CLINICAL TRIAL: NCT04100824
Title: Stellate Ganglion Block as Adjuvant Therapy to ca Channel Blocker in Prevention of Cerebrovascular Spasm in Traumatic Subarachnoid Hemorrhage
Brief Title: Stellate Ganglion Block as Adjuvant Therapy to ca Channel Blocker
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, m mostfa youssef mekky, Lecturer assistant, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: stellate ganglion block
Record Dates: First submitted 2019-09-19; First posted 2019-09-24 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Nimodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine 0.5% (Experimental): patient will take stellate ganglion block 10 ml bupivacaine 0.5% and nimodipine
  Interventions: Procedure: stellate ganglion block by transcranial doppler; Drug: Nimodipine
- Nimodipine (Active Comparator): patient will take nimodipine 60 mg every 4 h.
  Interventions: Drug: Nimodipine

INTERVENTIONS:
Procedure: stellate ganglion block by transcranial doppler — stellate ganglion block is a block of sympathetic ganglion
  Arms: Bupivacaine 0.5%
Drug: Nimodipine — Nimodipine 60mg every 4h

SUMMARY:
Aim of work:

To evaluate the effect of stellate ganglion block in prevention of cerebrovascular spasm in traumatic subarachnoid hemorrhage Primary outcome: Asses changes of cerebral blood flow velocity by Trans cranial Doppler.

Secondary outcome: Asses changes in clinical status

DETAILED DESCRIPTION:
A subarachnoid hemorrhage is a relatively uncommon type of stroke incidence and impact of traumatic brain injury hemorrhage (aSAH) has been extensively studied; less is (TBI) within the general population have increased known regarding the epidemiology of posttraumatic passover the past few years . It accounts for about 1 in 20 (5%) of all strokes. In contrast to common types of stroke, subarachnoid hemorrhage often occurs at a relatively young age half the patients are younger than 60 years. The outcome of patients after subarachnoid hemorrhage is generally poor. One of the causes of poor outcome is due to spasm and lack of blood supply to brain this occurs four to ten days after the hemorrhage.

Calcium antagonists as nimodipine are a type of drug that block calcium channels in cells and are often used for the treatment of high blood pressure. They have also been shown to counteract the narrowing of blood vessels after subarachnoid hemorrhage. Nimodipine is a dihydropyridine agent that blocks voltage-gated calcium channels and has a dilatory effect on arterial smooth muscle. It is the only FDA-approved agent for vasospasm with a half-life of about 9 h . Its beneficial effect on CVS derives most likely from its neuroprotective properties compared to arterial smooth muscle cell relaxation . The investigators can give nimodipine in several way as oral or IV and intrathecal .

Stellate ganglion block (SGB) has an established use in treating patients with disorders mediated by the sympathetic nervous system in which pain and/or circulatory insufficiency are predominant symptoms. These disorders include Atypical angina , post-herpetic neuralgia and complex regional pain syndromes, such as reflex sympathetic dystrophy .In addition, SGB has also been used, albeit somewhat controversially, in management of traumatic brain edema, schizophrenia, and complicated cervical migraine. However, the use of cervical sympathetic block has been described in reversing delayed ischemic neurologic deficit following aneurysmal subarachnoid hemorrhage.

The cerebral blood vessels, in particular the pia vessels, have a dense non-adrenergic sympathetic nerve supply that originates mainly in the cervical ganglia and accompanies the carotid artery to project into the ipsilateral hemisphere. There is controversy over the physiological significance of sympathetic innervation of the cerebral vasculature and the effect of SGB on it.The intracerebral vessels constrict in response to cervical sympathetic stimulation and dilate when these fibers are interrupted. The release and re-uptake of neurotransmitters, such as bradykinin, which is released during injury, can be prevented by sympathectomy. A recent report has suggested that cervical sympathetic block may be beneficial in patients with subarachnoid haemorrhage and that SGB may have therapeutic value in relieving cerebral vasospasm in certain neurological conditions. Anecdotal mention of SGB in some recent literature encourages the debate on its role as an adjunct to standard therapy for cerebral vasospasm, albeit, with a strong need for further evaluation

ELIGIBILITY:
Inclusion Criteria:

1. ASA: I, II
2. Head trauma
3. Hemodynamically stable patient
4. Mechanically ventilated or not
5. SAH diagnosed by CT brain

Exclusion Criteria:

1. relative refusal.
2. allergy to local anesthetic.
3. Any coagulation disorder.
4. Any vascular disease.
5. Penetrating head trauma.
6. Poly traumatized patient.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-11 (Actual); Primary Completion 2022-12-11 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
cerebral blood flow velocity | From 10 minutes to 24 hour after block
  Asses changes of cerebral blood flow velocity by Trans cranial Doppler

SECONDARY OUTCOMES:
clinical status | Over 10 days
  Asses changes in clinical status by galsco coma scale

CONTACTS AND LOCATIONS:
Locations (1):
- ِAssiut University Hospital, Asyut, Egypt